CLINICAL TRIAL: NCT00106041
Title: Randomized Trial of Care Management to Improve End of Life Care
Brief Title: Study to Improve Care for Veterans During Serious Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 02-294
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2012-09

CONDITIONS: Palliative Care
Keywords: end of life care; evaluation studies; quality of death and dying; palliative care; coordination of care; satisfaction with care; healthcare cost; utilization of healthcare resources; caregivers; veterans

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Palliative Care Nurse Case Management
  Interventions: Behavioral: Veterans Integrated Palliative Care Nurse Case Manager

INTERVENTIONS:
Behavioral: Veterans Integrated Palliative Care Nurse Case Manager — Palliative Care nurse case management

SUMMARY:
Improving end-of-life care is of critical importance to the VA as it faces an increasingly aging and dying veteran population. Previous work within and outside of the VA has demonstrated serious deficiencies in the quality of care delivered near the end of life. Moreover, veterans in the VA system suffer from a higher rate of chronic and life-limiting illnesses and decrements in health-related quality of life compared with the age-matched controls. In FY2000 approximately 104,000 enrolled veterans died in the U.S. including 27,200 that died as inpatients in VA acute or chronic care medical wards. The care model on which the proposed study is based is theoretically sound and has been piloted in a study that suggested its use can help the VA achieve substantial quality improvement at reduced costs.

DETAILED DESCRIPTION:
Background / Rationale: Improving end-of-life care is of critical importance to the VA as it faces an increasingly aging and dying veteran population. In FY2000 approximately 104,000 enrolled veterans died in the U.S. including 27,200 that died as inpatients in VA acute or chronic care medical wards. Previous work within and outside of the VA has identified serious deficiencies in the quality of care delivered near the end of life. A pilot program of a collaborative care intervention in patients with advanced illness suggests that palliative care management may lead to improvements in processes and outcomes of care at reduced costs.

Objective(s): The purpose of this project is to test the effectiveness of a chronic illness model-based palliative care intervention that utilizes prognosis-based palliative care evaluation and longitudinal nurse care management on the processes and outcomes of end-of-life care at one VA medical center.

Methods: The study uses a randomized, controlled design. All patients admitted to the inpatient medical service during the enrollment period are screened for survival prognosis by their admitting resident physician. Patients estimated to have at least a 25% risk of dying over the following year and who meet other basic inclusion criteria are invited to participate. Consenting patients are randomized to intervention or usual care. The intervention entails initial palliative evaluation followed by nurse care management designed to promote informed goal-setting, symptom management, psycho/socio/spiritual support, and family support. Data collection activities include patient and caregiver surveys, chart reviews, and reviews of administrative databases. Primary study outcomes include caregiver-rated quality of death and dying, hospital-based resource use, and costs; secondary outcomes include patient quality of life, satisfaction with care, continuity and coordination of care, and patient self-determination

Status: Enrollment and follow up of veterans/patients in the study is complete. Follow up with the caregivers of patients who died is ongoing and projected to end in February 2008. Subject enrollment began on 08/04/04 and target enrollment of 400 patients was reached in November 2006. Of the 1354 non-duplicated patients admitted to the hospital and prognostically eligible for the study, 795 (59%) were excluded; 400 (30%) were enrolled; 142(10%) refused; and 17 (1%) were missed or did not respond to recruitment efforts. To date, 257 of 400 enrolled veterans (64%) have died and 152 after-death interviews have been conducted with caregivers.

Impact: If shown to be effective, the palliative care program tested in this study will be the first of its type to demonstrate success in a controlled trial, and it will be ready for larger-scale implementation studies that will inform models of end-of-life care delivery both within and outside of the VA. Administrators at VAs nationwide, including chiefs of service, chiefs of staff, hospital directors, and VISN directors will be able to use the plans and protocols developed in this project to develop programs at their own institutions. Nurses, generalist physicians, and specialists can gain important insights about the special needs of seriously ill patients and the role of care systems in delivering high-quality end of life care. Finally, the project has immediate relevance to the healthcare system at large, as it struggles to find effective end-of-life care delivery models.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to the hospital's general medicine service and estimated to have at least a 25% risk of dying over the following year.

Exclusion Criteria:

* Inability to pass cognitive screen
* Homelessness
* No telephone
* Admission from or discharge to a nursing home or hospice care
* Enrollment in another healthcare program or study that duplicates services of this study
* Receives most healthcare/primary healthcare services outside the VA GLA catchment area
* Does not speak English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Healthcare expenditures including inpatient, ICU, outpatient, pharmacy and total costs; utilization of healthcare resources; and quality of death and dying experience. Includes expenditures time of study enrollment until patient's death. | We will be tracking resource use until the death of the patient or the conclusion of the study, whichever comes first. Quality of the death and dying experience will be assessed within 90 days of death

SECONDARY OUTCOMES:
Satisfaction with care, quality of care, symptom management, understanding of illness, continuity and coordination of care, end-of-life care preferences, advance care planning, and treatments. | This will be assessed during the first year of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E. Rosenfeld, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Result] Wagner GJ, Riopelle D, Steckart J, Lorenz KA, Rosenfeld KE. Provider communication and patient understanding of life-limiting illness and their relationship to patient communication of treatment preferences. J Pain Symptom Manage. 2010 Mar;39(3):527-34. doi: 10.1016/j.jpainsymman.2009.07.012. Epub 2010 Feb 19. PMID 20171827
- [Result] Seow H, Snyder CF, Shugarman LR, Mularski RA, Kutner JS, Lorenz KA, Wu AW, Dy SM. Developing quality indicators for cancer end-of-life care: proceedings from a national symposium. Cancer. 2009 Sep 1;115(17):3820-9. doi: 10.1002/cncr.24439. PMID 19514090
- [Result] Goebel JR, Doering LV, Lorenz KA, Maliski SL, Nyamathi AM, Evangelista LS. Caring for special populations: total pain theory in advanced heart failure: applications to research and practice. Nurs Forum. 2009 Jul-Sep;44(3):175-85. doi: 10.1111/j.1744-6198.2009.00140.x. PMID 19691653
- [Result] Fromme EK, Hughes MT, Brokaw FC, Rosenfeld KE, Arnold RM. Update in palliative medicine 2008. Journal of palliative medicine. 2008 Jun 1; 11(5):769-75.
- [Result] Casarett D, Pickard A, Amos Bailey F, Ritchie C, Furman C, Rosenfeld K, Shreve S, Shea JA. Important aspects of end-of-life care among veterans: implications for measurement and quality improvement. J Pain Symptom Manage. 2008 Feb;35(2):115-25. doi: 10.1016/j.jpainsymman.2007.03.008. Epub 2007 Nov 28. PMID 18053680
- [Result] Lorenz KA, Lynn J, Dy SM, Shugarman LR, Wilkinson A, Mularski RA, Morton SC, Hughes RG, Hilton LK, Maglione M, Rhodes SL, Rolon C, Sun VC, Shekelle PG. Evidence for improving palliative care at the end of life: a systematic review. Ann Intern Med. 2008 Jan 15;148(2):147-59. doi: 10.7326/0003-4819-148-2-200801150-00010. PMID 18195339
- [Result] Lorenz KA, Rosenfeld K, Wenger N. Quality indicators for palliative and end-of-life care in vulnerable elders. J Am Geriatr Soc. 2007 Oct;55 Suppl 2:S318-26. doi: 10.1111/j.1532-5415.2007.01338.x. No abstract available. PMID 17910553
- [Result] Chang VT, Sorger B, Rosenfeld KE, Lorenz KA, Bailey AF, Bui T, Weinberger L, Montagnini M. Pain and palliative medicine. J Rehabil Res Dev. 2007;44(2):279-94. doi: 10.1682/jrrd.2006.06.0067. PMID 17551879
- [Result] Krouse RS, Mohler MJ, Wendel CS, Grant M, Baldwin CM, Rawl SM, McCorkle R, Rosenfeld KE, Ko CY, Schmidt CM, Coons SJ. The VA Ostomy Health-Related Quality of Life Study: objectives, methods, and patient sample. Curr Med Res Opin. 2006 Apr;22(4):781-91. doi: 10.1185/030079906X96380. PMID 16684439